CLINICAL TRIAL: NCT06558617
Title: Evaluating SARC-F, SARC-CalF, and Calf Circumference as Diagnostic Tools for Sarcopenia in Thai Older Adults: Results From a Nationwide Study
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Panai Laohaprasitiporn, MD, Assistant Professor, Siriraj Hospital
Other Study IDs: COA-023/2024
Record Dates: First submitted 2024-08-10; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia; Diagnosis
Keywords: sarcopenia; calf circumference; SARC-F questionnaire; diagnostic accuracy; elderly
MeSH Terms: conditions — Sarcopenia; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thai community-dwelling older adults
  Interventions: Diagnostic Test: SARC-F Questionnaire; Diagnostic Test: Calf Circumference Measurement; Diagnostic Test: SARC-CalF Questionnaire

INTERVENTIONS:
Diagnostic Test: SARC-F Questionnaire — The SARC-F scale consists of five components: strength, walking assistance, rising from a chair, stair climbing, and falls. These elements were selected to reflect changes in health status related to the effects of sarcopenia. Scores on the SARC-F scale range from 0 to 10, composed of five domains, assesses strength, walking assistance, raising from a chair, stair climbing and falls. Each domain score ranges from 0-2. A SARC-F score of ≥4 was considered abnormal. The Thai-version SARC-F questionnaire has been validated in Thai older adults.
Diagnostic Test: Calf Circumference Measurement — Calf circumference was measured using a nonelastic tape measure while the participant was standing with relaxed legs. The tape was placed snugly and flat around the widest part of the calf, parallel to the floor. According to the AWGS 2019 criteria, calf circumferences were considered abnormal if they were less than 34 cm for males and less than 33 cm for females.
Diagnostic Test: SARC-CalF Questionnaire — This questionnaire integrates the SARC-F and calf circumference as a trigger for case finding. If the calf circumference is below the cut-off value, 10 points are added to the SARC-F score for evaluation. The SARC-CalF score ranges from 0 to 20, with a score of ≥11 considered abnormal for sarcopenia screening.

SUMMARY:
As the elderly population grows, musculoskeletal disorders, including sarcopenia, have become a critical area of study due to their association with falls and fractures. Sarcopenia, characterized by decreased muscle mass, is prevalent among older adults and poses a significant risk for falls. This study aimed to assess the effectiveness of the SARC-F and SARC-CalF questionnaires, along with calf circumference measurements, in screening for sarcopenia among Thai community-dwelling older adults, following the Asian Working Group on Sarcopenia (AWGS) 2019 criteria.

DETAILED DESCRIPTION:
The data utilized in this analysis were derived from the Thai Musculoskeletal Diseases Nationwide Study. This cross-sectional study targeted Thai adults aged 60 years and older, conducted between March 2021 and August 2022. Participants were sampled using a multi-level sampling technique to ensure representativeness from community-dwelling older adults across 12 provinces, encompassing Thailand's six primary geographical regions.

Participants were evaluated for possible sarcopenia or sarcopenia, according to AWGS 2019 criteria, by using SARC-F questionnaire, calf circumference measurement, SARC-CalF questionnaire, and appendicular skeletal muscle mass (ASM).

ELIGIBILITY:
Inclusion Criteria:

* Thai adults aged 60 years and older

Exclusion Criteria:

* missing data on SARC-F, SARC-CalF, and calf circumference
* unable to walk independently
* bedridden individuals
* neuromuscular disorders or severe comorbidities that could impair their ability to perform performance-based tests

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older Thai adults living at that area for at least 1 year
Sampling Method: Probability Sample
Enrollment: 2543 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass (ASM) | up to 4 weeks
  To assess appendicular skeletal muscle mass (ASM), we used the Tanita RD-545, a dual-frequency bioelectrical impedance analysis (BIA) device (Tanita Corporation, Tokyo, Japan). Previous studies have demonstrated that this BIA method is reliable and comparable to dual-energy X-ray absorptiometry (DXA) for diagnosing sarcopenia in Thai elderly adults. The appendicular skeletal muscle mass index (ASMI) was calculated by dividing the ASM by the square of the height. According to the 2019 criteria of the AWGS, low muscle mass is defined as <7.0 kg/m² for men and <5.7 kg/m² for women.
Handgrip strength | up to 4 weeks
  Participants were asked to squeeze a digital Smedley spring hand dynamometer (Takei 5401 Digital Dynamometer; Takei, Tokyo, Japan) with maximum effort while standing with fully extended arms at their sides. The grip size was adjusted for each participant's hand size, and 2 or 3 trials were performed, with the highest output value recorded. Handgrip strengths < 28 kg in males and < 18 kg in females were classified as low muscle strength, per the AWGS 2019 criteria.
5-time sit-to-stand test (5TSTS) | up to 4 weeks
  Participants were directed to sit upright on armless chairs with their backs supported firmly by the backrest. They were then instructed to stand up as quickly as possible for 5 repetitions with their arms crossed, trunk upright, and hips and knees fully extended. The time taken by each participant to complete the test from the initial sitting to the fifth sitting was recorded. The test is considered abnormal if it takes equal or more than 12 seconds to complete the task.

CONTACTS AND LOCATIONS:
Overall Officials: Apichat Asavamongkolkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanitcharoenkul E, Unnanuntana A, Chotiyarnwong P, Adulkasem N, Asavamongkolkul A, Laohaprasitiporn P. Evaluating SARC-F, SARC-CalF, and calf circumference as diagnostic tools for sarcopenia in Thai older adults: results from a nationwide study. BMC Geriatr. 2024 Dec 28;24(1):1043. doi: 10.1186/s12877-024-05637-3. PMID 39732657